CLINICAL TRIAL: NCT02180022
Title: Effect of Onion Peel Extract on Endothelial Function and Endothelial Progenitor Cells in Overweight and Obese Subjects
Brief Title: Effects of Onion Peel Extract on Endothelial Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Kyunghee University (Other)
Responsible Party: Principal Investigator, Weon Kim, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Onion-EPC; Seoul, Korea (Other Grant/Funding Number: No. 1111473)
Record Dates: First submitted 2014-06-28; First posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Healthy; Overweight; Obese
Keywords: Quercetin; Endothelial function; Onion peel extract; volunteers
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients treated with placebo for 12 weeks
  Interventions: Drug: Placebo
- Onion peel extract (Experimental): Patients treated with onion peel extract for 14 days
  Interventions: Drug: Onion peel extract

INTERVENTIONS:
Drug: Placebo — After randomization, placebo was treated for 12 weeks
  Arms: Placebo
Drug: Onion peel extract — After randomization, onion peel extract was treated for 12 weeks
  Other Names: OPE
  Arms: Onion peel extract

SUMMARY:
Acute or chronic intake of polyphenol-rich foods has been reported to improve endothelial function. Quercetin, found abundantly in onion, is a potent antioxidant flavonoid. This study was designed to investigate whether consumption of onion peel extract (OPE) improves endothelial function in healthy overweight and obese subjects.

DETAILED DESCRIPTION:
Epidemiological studies have shown a rapid increase in the prevalence of overweight and obesity, not only in adults but also in children and adolescents, thus increasing the risk of early development of cardiovascular disease (CVD). Quercetin, found abundantly in onion, prevents the induction of endothelial dysfunction, superoxide production, and overexpression by angiotensin II in the rat aorta. Furthermore, in our previous study we showed that supplementation with quercetin-rich onion peel extract (OPE) influenced adipokine expression, thus addressing its modulatory effect on obesity-induced inflammation, and improved insulin resistance by alleviating the metabolic dysregulation of free fatty acids, suppressing oxidative stress, upregulating glucose uptake, and downregulating inflammatory gene expression. But there are limited studies on the relationship between quercetin supplementation and endothelial dysfunction in humans.

ELIGIBILITY:
Inclusion Criteria:

* age 20 to 60 years
* BMI >23 kg/m2
* abdominal circumference > 90 cm in males or >85 cm in females

Exclusion Criteria:

* hypertension (>140/90 mmHg),
* diabetes
* any cardiovascular disease,
* kidney disease,
* thyroid disease
* cerebrovascular disease
* liver disease (bilirubin level >2 mg/dl)
* pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The difference of endothelial function | 12 weeks after study drug treatment
  The difference of forearm FMD (flow meidated dilation) achieved following study drug treatment

SECONDARY OUTCOMES:
The difference of EPC (endothelial progenitor cell) counts | 12 weeks after study drugs treatment
  After appropriate gating based on low cytoplasmic granularity and low expression of CD45, CD34+VEGFR2+ cells were counted and expressed as the number of cells/106 total events or number of cells/100 µL of blood.

OTHER OUTCOMES:
The composite measure of change of blood pressure, heart rate, body weight and blood chemistry | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Weon Kim, MD, PhD, Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea